CLINICAL TRIAL: NCT06327971
Title: Enhanced Outcome Prediction in Cutaneous Squamous Cell Carcinoma Using Deep-learning and Computational Histopathology
Status: Active, not recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 0000
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Squamous Cell Carcinoma of the Skin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate a deep-learning model trained on computational histopathology for predicting outcomes in cutaneous squamous cell carcinoma

ELIGIBILITY:
Histologically-confirmed diagnosis of primary cutaneous squamous cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Metastasis | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, United Kingdom